CLINICAL TRIAL: NCT01636973
Title: Effects of Humidified Ventilation on Arterial Oxygenation and Respiratory Mechanics During One Lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double
Other Study IDs: 1-2011-0027
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Lung Cancer
Keywords: Lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaporizing humidifier (Experimental): Vaporizing humidifier applying during one-lung ventilation
  Interventions: Procedure: Vaporizing humidifier

INTERVENTIONS:
Procedure: Vaporizing humidifier — Vaporizing humidifier applying during one-lung ventilation

SUMMARY:
A continuous loss of moisture and heat occurs during mechanical ventilation and prediposes patients to airway damage. Vaporizing humidifier has known to be advantages of improvement of oxygenation and protection of airway damage. However, there is a lack of study about the effect of humidified ventilation on oxygenation and respiratory mechanics during one-lung ventilation. We therefore invesgate that the effect of humidified ventilation on oxygenation and respiratory mechanics during one-lung ventilation .

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status class I,II
* Unilateral lung lobectomy
* Use of one-lung ventilation

Exclusion Criteria:

* COPD
* CAOD
* Unstable cardiovascular status
* Peak inspiratory pressure > 30 mmHg

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
arterial oxygenation | T1(10min before one-lung ventilation),T2(30min after one-lung ventilation),T3(60min), T4(10min after two lung ventilation)
  T1,T2,T3,T4: all measurement in lateral position, T1-arterial oxygenation(PaO2), T2-arterial oxygenation(PaO2),T3-arterial oxygenation(PaO2),T4-arterial oxygenation(PaO2)

SECONDARY OUTCOMES:
Respiratory dynamic parameters | T1,T2,T3,T4 (same as 'primary outcome measure')
  T1,T2,T3,T4: T1-respiratory dynamic parameters, T2-respiratory dynamic parameters, T3-respiratory dynamic parameters, T4-respiratory dynamic parameters

CONTACTS AND LOCATIONS:
Overall Officials: Young Jun Oh, M.D.,PhD., Study Chair — Yonsei University
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea